CLINICAL TRIAL: NCT05375123
Title: Reference Range for Tissue Motion Tracking of Mitral Annulus Displacement in Chinese Han Singleton Pregnancies: a Prospective, Multicenter, Clinical Trial
Brief Title: Reference Range for Tissue Motion Tracking of Mitral Annulus Displacement in Chinese Han Singleton Pregnancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Ma, Chief of Cardiovascular Ultrasound, First Hospital of China Medical University
Other Study IDs: REVAW-TMAD-01
Record Dates: First submitted 2022-04-29; First posted 2022-05-16 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Pregnancy
Keywords: Pregnancy; Left Ventricular Systolic Function; Tissue Motion Tracking of Mitral Annular Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trial group: A total of 660 singleton pregnant women in the first trimester (gestational age of 6-13 weeks + 6 days), who had normal results in various examinations and experienced regular obstetric examinations throughout the pregnancy, were selected from the obstetric outpatients in 33 centers, with 20 cases in each center.
  Interventions: Device: Ultrasound image acquisition

INTERVENTIONS:
Device: Ultrasound image acquisition — Echocardiography: left ventricular systolic function of all participants were measured by tissue motion tracking of mitral annular displacement using PHILIPS.
  Time points for heart image acquisition in pregnant women: As per the Guidelines for Pre-pregnancy and Pregnancy Health Care (2018) formulated by the Obstetrics Group of the Gynecology Branch of the Chinese Medical Association, a total of six echocardiographic examinations will be performed in the first trimester (11-14 weeks of gestation), the second trimester (20-24 weeks of gestation), the third trimester (29-32 weeks of gestation), prenatal term (37-41 weeks of gestation), 6 weeks and 3-6 months after delivery.
  Time points for fetal heart image acquisition: Fetal heart images will be collected in the second trimester (20 to 24 weeks of gestation).

SUMMARY:
The First Affiliated Hospital of China Medical University initiated a multi-center study on the reference range of tissue motion tracking of mitral annulus displacement in Chinese Han singleton pregnancies to determine the reference range of tissue motion annular displacement (TMAD) in the pregnant population and to promote the clinical application of TMAD in the pregnant population, thereby offering new insights into the early evaluation and early diagnosis for cardiac function in the pregnant population.

DETAILED DESCRIPTION:
During normal pregnancy, the cardiovascular system of pregnant women will undergo significant adaptive changes in response to the growth of the uterus, fetus and placenta. Cardiac output and plasma volume will increase by 40% to 50% compared with non-pregnancy. The heart rate continues to increase, while the blood pressure decreases in the first and second trimesters and increases in the third trimester. The heart structure of pregnant women also remodels during pregnancy and the inner diameter of the cardiac cavity and myocardial mass increase. The above changes usually return to pre-pregnancy levels within 3-6 months after delivery. Pregnancy can change hemodynamics and cardiac structure, thereby causing corresponding changes in maternal cardiac function. Adaptive changes in maternal cardiac function can be reflected through an accurate and rapid evaluation. Changes in maternal cardiac function can be continuously observed and analyzed during pregnancy and after delivery to uncover the changing law of maternal cardiac function.

In addition, the incidence of cardiovascular disease in pregnancy is 1-4% worldwide, and about 15% of maternal deaths are caused by complications related to cardiovascular diseases during pregnancy. In China, the proportion of maternal deaths caused by cardiovascular diseases during pregnancy is increasing yearly and cardiovascular diseases during pregnancy have become the primary cause of death for critically ill pregnant women. Previous studies have shown that common complications during pregnancy, such as gestational hypertension and diabetes, can also alter maternal heart function. Therefore, early detection of changes in left ventricular systolic function of pregnant women during pregnancy and after childbirth, timely treatment and early evaluation of treatment efficacy can greatly reduce their mortality.

The Simpson's biplane method is currently used to measure left ventricular ejection fraction for clinical evaluation of left ventricular systolic function, which is especially available for patients without left ventricular geometric deformation. However, left ventricular ejection fraction cannot be sensitive to early changes in cardiac function. In recent years, two-dimensional longitudinal strain has been included for evaluating left ventricular systolic function. Myocardial longitudinal motion is responsible for maintaining 70% of normal cardiac function. Researchers believe that this method can sensitively detect early changes in left ventricular systolic function. However, the above two methods have high requirements on the quality of ultrasound images, which can clearly display the endocardium and epicardium based on good sound-transmitting conditions and good image quality. However, the image quality of pregnant women is often poor, so there is a decline in the detection accuracy.

Previous studies have shown that TMAD is independent of image quality and can effectively evaluate left ventricular systolic function and is an effective supplement to left ventricular ejection fraction and the overall longitudinal strain of the left ventricle. TMAD is a new technique for quantitative analysis of mitral annulus motion parameters. Three observation points are set on the septal side, lateral side and apex of the mitral annulus in the apical four-chamber view. The movement of the mitral annulus relative to the apex will be detected to obtain the lateral displacement of the mitral annulus septum (TMAD sep), the lateral displacement of the mitral annulus (TMAD lat), the mean displacement (TMADmid), and the mean displacement rate (TMADmidpt%). The left ventricular longitudinal systolic function will be then evaluated. TMAD only requires image acquisition from three sites and has low requirements on the quality of ultrasound images. Therefore, this measurement is simple, accurate and highly repeatable.

However, the TMAD reference value of normal healthy adults cannot be directly applied to pregnant women due to the hemodynamic changes during pregnancy. It is still necessary to establish the reference value of TMAD in pregnant women and explore its changes with gestational age, so as to provide simple, fast, accurate ultrasound parameters that do not depend on image quality for the evaluation of cardiac function during pregnancy.

The purpose of this study is to establish the reference range of TMAD parameters in Chinese Han singleton pregnancies in different pregnancy periods and early postpartum period and to explore the influencing factors of TMAD in singleton pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy;
* Han nationality;
* 18-45 years old;
* Basal body mass index before pregnancy < 30 kg/m2;
* Normal blood pressure (139-90/89-60 mmHg);
* No history of cardiovascular and respiratory diseases;
* No abnormal findings in the physical examination of the cardiovascular and respiratory systems;
* Normal results in blood, urine, fasting blood glucose, blood lipids, liver and kidney function, thyroid function and electrocardiogram;
* Echocardiography shows normal cardiac function with no structural heart diseases;
* No use of medications that affect the cardiovascular system.

Exclusion Criteria:

* Multiple pregnancy;
* Anemia (hemoglobin < 90 g/L);
* Other serious diseases of the immune, respiratory, digestive, nervous, urinary, blood, endocrine and other systems;
* Tumors;
* The poor quality of ultrasound images cannot meet the requirements of parameter measurement and analysis.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: A total of 660 singleton pregnant women in the first trimester, who had normal results in various examinations and experienced regular obstetric examinations throughout the pregnancy, were selected from the obstetric outpatients in 33 centers, with 20 cases in each center.
Sampling Method: Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of left ventricular systolic function in Chinese Han singleton pregnancies using the TMAD method | From 11 weeks of gestation to 3-6 months postpartum
  To establish the reference range of TMADmid and TMADmidpt% in Chinese Han singleton pregnancies using the TMAD method.

SECONDARY OUTCOMES:
Measurement of left ventricular systolic function using the Simpson's biplane method | From 11 weeks of gestation to 3-6 months postpartum
  Measurement of left ventricular ejection fraction measured by the Simpson's biplane method is a clinical standard

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Ma, MD, Principal Investigator — First Hospital of China Medical University
Locations (33):
- China (33):
  - Chongqing Fifth People's Hospital, Chongqing, Chongqing Municipality
  - Chongqing Banan District People's Hospital, Chongqing, Chongqing Municipality
  - Chongqing Qianjiang District Central Hospital, Chongqing, Chongqing Municipality
  - Maternity and Child Care Centers of Fujian Province, Fuzhou, Fujian
  - Hainan Women and Children's Medical Center, Haikou, Hainan
  - Jiamusi Central Hospital, Jiamusi, Heilongjiang
  - Nanyang First People's Hospital, Nanyang, Henan
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Center Hospital of Wuhan, Wuhan, Hubei
  - Maternal and Child Health Care Hospital Hubei, Wuhan, Hubei
  - Jilin Provincial Women and Children Health Hospital, Changchun, Jilin
  - Jilin People's Hospital, Jilin, Jilin
  - Jilin Central General Hospital, Jilin, Jilin
  - Siping Women and Infants Hospital, Siping, Jilin
  - Yanji Maternal and Infant Hospital, Yanji, Jilin
  - Dalian Friendship Hospital, Dalian, Liaoning
  - Dalian Municipal Women and Children's Medical Center, Dalian, Liaoning
  - Women And Children's Hospital of Jinzhou, Jinzhou, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shenyang Maternity And Child Health Hospital, Shenyang, Liaoning
  - the First Hospital of China Medical Univeristy, Shenyang, Liaoning
  - Tieling Women's And Children's Hospital, Tieling, Liaoning
  - Ningxia Maternal And Child Health Care Hospital, Yinchuan, Ningxia
  - Qinghai Provincial Maternal and Child Health Hospital, Xining, Qinghai
  - ShaanXi Province People's Hospital, Xi'an, Shaanxi
  - Heze Municipal Hospital, Heze, Shandong
  - Shandong Maternal and Child Health Hospital, Jinan, Shandong
  - Weifang Maternal and Child Health Hospital, Weifang, Shandong
  - ZiBo Central Hospital, Zibo, Shandong
  - Panzhihua Maternal and Child Hospital, Panzhihua, Sichuan
  - Yaan People's Hospital, Ya'an, Sichuan
  - Yunnan Maternal And Child Health Care Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided